CLINICAL TRIAL: NCT02780921
Title: Effect of Prehabilitation in Gastroesophageal Adenocarcinoma: Study Protocol of a Multicentric, Randomised Control Trial
Acronym: PREHAB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0263; 2015-A01733-46 (Registry Identifier: 2015-A01733-46)
Record Dates: First submitted 2016-04-28; First posted 2016-05-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Oesophageal Cancer; Gastric Cancer
Keywords: Prehabilitation; Oesophageal cancer; Gastric cancer; Fitness; Preconditionning; two parallel arms
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Preoperative Exercise; Nutritional Support

ARMS (2):
- Prehab Group (Experimental): In the experimental group (Prehab group) compared to the control group, the main objective will be to demonstrate an improvement of the percentage of patients reaching the complete oncological treatment fixed in a multidisciplinary tumour board
  Interventions: Procedure: prehabilitation
- control group (Other): The control group will be treated according to conventional care; will not receive any specific intervention before surgery except nutritional support and physiotherapy at the surgeon's discretion
  Interventions: Other: nutritional support

INTERVENTIONS:
Procedure: prehabilitation
  Arms: Prehab Group
Other: nutritional support
  Arms: control group

SUMMARY:
Perioperative chemotherapy is the gold standard treatment in the resectable and advanced gastroesophageal adenocarcinoma. The efficacy of this strategy has been demonstrated in two randomized studies (1,2). It reduces tumour size before surgery, treats micrometastases and evaluates chemosensitivity. Disease free and overall survival rates were significantly improved with perioperative chemotherapy compared to surgery alone. However, the limitation of these studies is that among all patients requiring chemotherapy, almost 70% of patients will not have the complete sequence. This sequence is defined by the administration of 2 to 4 cycles before and 2 to 4 cycles after the surgery, according to the protocol. The major cause of absence or impossibility of realization of postoperative chemotherapy was the presence of postoperative complication, postoperative serious asthenia and impaired nutritional and physical status (1,2). Poor physical condition assessed by cardiopulmonary exercise testing, reflecting a reduced physiological reserve, is predictive of postoperative complications (3,4). A physical training, even during a short period and on a various population, is beneficial in improving physical condition, cardiopulmonary function and muscular mass of the patient (5-8). A prehabilitation over a 6 week period between surgical consultation and surgery decreases postoperative morbidity and the hospital stay in cardiovascular surgery but no study has ever been performed in the gastric or oesophageal cancer (7,9).

Prehabilitation revolves around three axes: 1) a physical training based on initial cardiopulmonary exercise testing (VO2peak, anaerobic threshold (AT) and 6-min walk test (6MWT)), 3 times by week, supervised by a physical therapist 2) a nutritional care to ensure the compliance of the nutrition program and adapt the nutritional management based on protein and energy needs and on the level of spontaneous oral intake and 2) a psychological treatment by a psychologist to reduce preoperative anxiety. To our knowledge, no study ever focused on the gastroesophageal cancer. The benefit of prehabilitation in this cancer may be particularly important because 1) this surgery is associated with a high postoperative morbidity (40%, especially respiratory) and mortality (5%) 2) the physical and nutritional status of these patients is often precarious (cancer cachexia, gastroesophageal obstruction), and 3) the need to preoperative chemotherapy declines physical reserves and is associated with a lengthening of the time between consultation and surgery of more than 3 months (10). Also, the investigators hypothesize that with a physical training, a personalized nutritional support and a psychologist management may decrease postoperative complications, increase postoperative nutritional status and so, would allow for more patients to receive their full cancer treatment. The aim of this study was to evaluate, in gastroesophageal adenocarcinoma, the effect of prehabilitation compared to conventional care, the percentage of patients reaching the complete oncological treatment decided in a multidisciplinary tumour board.

DETAILED DESCRIPTION:
Interventions After the first visit with his surgeon, the patient will be presented at the multidisciplinary tumour board to validate the inclusion criteria and to schedule the number of cycles of pre- and postoperative chemotherapy. After this step, a second consultation with the surgeon will allow to verify all inclusion and exclusion criteria and perform the randomization. For the two groups, an initial (before chemotherapy) and final (one week before the surgery) evaluation will be performed. The evaluation includes cardiopulmonary exercise testing (VO2peak, AT and 6MWT), nutritional evaluation (albumin), bioelectric impedance analysis, evaluation of physical activity and ingesta, evaluation of the level of depressive symptoms and anxiety with the HADS questionnaire and the quality of life (5Q-FD questionnaire).

Prehab group Exercise intervention: The total-body exercise will consist of up to 1 hour of supervised exercise for at least 3 days per week, for a total of 18 cycles, alternating between aerobic and resistance training. Exercise intensity will be prescribed based on the rate of the 6MWT, AT and VO2peak. The participant will exercise in the presence of the kinesiologist who will provide corrective feedback if necessary.

Nutrition intervention: Initially, a nutritionist will perform a medical and biological examination of the nutritional status to provide individualized care to each patient. Individual protein requirements will be calculated as 1.2 g of protein per kilogram of body weight (adjusted body weight was used for obese patients), as per European Society for Clinical Nutrition and Metabolism (ESPEN) guidelines, regarding surgical patients (12). Patients will be asked to consume the protein supplement within one hour of their exercise regimen to capitalize on postexercise muscle protein synthesis (13). Then, a dietician will assess the compliance of the nutritional support at each cycle of chemotherapy and will adjust it if necessary. After the preoperative chemotherapy, a second evaluation by a nutritionist will be performed.

Psychologist intervention: Patients will receive up to a one hour visit with a trained psychologist who will provide techniques aiming to reducing anxiety, such as relaxation exercises based on imagery and visualization, together with breathing exercises. Each patient will practice these exercises with the psychologist initially and at each cycle of chemotherapy and at home two to three times per week. The psychologist also provides suggestions on how to enhance and reinforce patients' motivation to comply with the exercise and nutritional aspects of the intervention.

Control group:

The control group will be treated according to conventional care; will not receive any specific intervention before surgery except nutritional support and physiotherapy at the surgeon's discretion.

ELIGIBILITY:
Inclusion Criteria:

> 18 years old.

* Patient who agreed to participate in the study
* Patient requiring surgical management for the cancer of the esophagus or stomach.
* Patient who have a standard perioperative chemotherapy:

For esophageal cancer: chemotherapy with 5-FU (or LV5-FU2) -platinum salts or Taxane-salt platinum salts, 2 to 4 cycles pre- and postoperatively.

For stomach cancer: Perioperative chemotherapy with Epirubicin and cisplatin-5-FU (ECF), Epirubicin-oxaliplatin-5FU (EOX) or 5-FU (or LV5FU) - platinum salts, 2 to 4 cycles.

* subscribe to the French national health insurance system and give their written consent.
* Patient speak and understand French.
* effective contraception for patients of childbearing age

Exclusion Criteria:

* Patient who for psychiatric social, family or geographical reasons, will not be able to be monitored and/or compliant with the requirements of the study.
* Patient requiring preoperative radio-chemotherapy. with any unbalanced progressive disease (hepatic failure, renal failure (creatinine clearance <30mL / min), respiratory failure, congestive heart failure, myocardial infarction in the last 6 months)
* Patient treated for another cancer within 5 years, except basal cell skin carcinoma or carcinoma in situ of the cervix.
* patient in legal incapacity (person deprived of liberty or under guardianship).
* cognitive disorders or major disability making it impossible to understand the study and sign the informed consent
* breastfeeding or pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
percentage of patients reaching the complete oncological treatment fixed in a multidisciplinary tumour board | at inclusion
  In the experimental group (Prehab group) compared to the control group, the main objective will be the percentage of patients reaching the complete oncological treatment fixed in a multidisciplinary tumour board.

SECONDARY OUTCOMES:
effect of the prehabilitation on the postoperative morbidity on the postoperative morbidity according Dindo-Clavien classification | at 3 months
  according Dindo-Clavien classification, a scale from 0 (no postoperative morbidity) to 5 (postoperative death)
evaluation of the effect of the prehabilitation on severe morbidity (Clavien >2) | at 3 months
  severe morbidity at 3 months (Clavien >2), defined by an interventional or surgical treatment
disease free survival (DFS) | at 3 and 5 years
  disease free survival (DFS), survival defined by the time in months before recurrence at 3- and 5-years after the end of the postoperative chemotherapy
overall survival (OS) | at 3 and 5 years
  overall survival (OS), defined by the time in months of the overall survival at 3- and 5 years after the end of the postoperative chemotherapy.
feasibility of the protocol | at inclusion
  feasibility of the protocol defined by the percentage of physical sessions realized on the eighteen proposed in the preoperative period
length (in days) of postoperative stay | at 3 months
difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) VO2 at the ventilatory threshold (ml.min-1.kg-1). | at 3 months
difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) value of VO2peak (ml.min-1.kg-1.). | at 3 months
difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) walking distance in 6 min (meters). | at 3 months
difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) weight (Kg) | at 3 months
difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) albuminemia (g/l) | at 3 months
evaluation on the score of HADS survey (Hospital anxiety and depression scale) | at 3 months
  difference between the initial (before preoperative chemotherapy) and final (after preoperative chemotherapy) evaluation on the score of HADS survey (Hospital anxiety and depression scale) to assess the anxiety and depression from a survey with 14 questions.
quality of life | at 3 months
  difference of the score between the initial evaluation (before preoperative chemotherapy) and at 3-months after the surgery of the quality of life defined by the EQ-5D survey.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Le Roy B, Pereira B, Bouteloup C, Costes F, Richard R, Selvy M, Petorin C, Gagniere J, Futier E, Slim K, Meunier B, Mabrut JY, Mariette C, Pezet D. Effect of prehabilitation in gastro-oesophageal adenocarcinoma: study protocol of a multicentric, randomised, control trial-the PREHAB study. BMJ Open. 2016 Dec 7;6(12):e012876. doi: 10.1136/bmjopen-2016-012876. PMID 27927660